CLINICAL TRIAL: NCT04966754
Title: Data Driven Behavior Intervention and Medical Outcome Evaluation of Patients' Comprehensive Monitoring
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Peking University (Other); Guangdong Provincial People's Hospital (Other); Guangzhou Huyun Hospital Management Co., Ltd (Unknown)
Responsible Party: Sponsor
Other Study IDs: JS-2898
Record Dates: First submitted 2021-07-08; First posted 2021-07-19 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Metabolic Syndrome; Metabolic Disturbance; Metabolic Complication; Infection; Obesity; Diabetes
Keywords: metabolic; diabetes; obesity; infection; complication
MeSH Terms: conditions — Metabolic Syndrome; Infections; Obesity; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
During the study, the resuscitation room, general wards and ICU were installed fixed or mobile acquisition devices in the resuscitation room, the emergency department of Peking Union Medical College Hospital, and the collection platform was set up. Patients with acute diseases (infection, diabetes complications, etc.) caused by metabolic syndrome (obesity, diabetes, etc.) were selected after informed consent. All medical intervention behaviors, relevant medical records and medical outcome records within the collection scope of the device platform were collected prospectively . And regular follow-up, guidance of patients with metabolic syndrome control, while collecting all the lifestyle characteristics of patients, some patients with metabolic cabin research, and observe the relevant medical outcomes. After that, all the collected data were coded, and the influence of all lifestyle and medical behavior interventions on patients' medical outcomes was studied by artificial intelligence method.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes and / or obesity (BMI>=28).
* Emergency room / emergency ward / EICU;
* Be able to understand and agree the research protocol and sign the informed consent

Exclusion Criteria:

* Pregnant women / lactation period;
* The estimated survival time was less than 1 year;
* Long term follow-up is not guaranteed;
* Failure to comply with the protocol or procedure;
* The collection of medical behavior data can not complete the de privacy or label after de privacy;
* Other researchers think that it is not suitable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metabolic syndrome (obesity, diabetes, etc.) cause acute disease attacks (infection, diabetes complications, etc.).
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-11-30 (Estimated)

PRIMARY OUTCOMES:
Rate of metabolic complications | 6 weeks
  Relapse of acute metabolic disease, stability of biochemical metabolic indexes (such as glycosylated hemoglobin, BMI)
Complication control | 3 weeks
  The occurrence of metabolic complications, infection and cardiovascular events
Rate of mortality | 6 months
  30-day and 90-day mortality. Death due to cardiovascualr complications

SECONDARY OUTCOMES:
Total cost of treatment | 3 weeks
  Length of stay, length of stay in ICU, ventilator usage time
Quality of life | 6 months
  Dynamic monitoring of quality of life through quality-of-life evaluation chart

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2021-07-06): https://cdn.clinicaltrials.gov/large-docs/54/NCT04966754/Prot_000.pdf